CLINICAL TRIAL: NCT04644653
Title: Steered t-PA Delivery for Thrombolysis Test Using Magnetic Swarming Nanorobots on Human Placenta as an ex Vivo Model of Human Cerebral Vascular System
Brief Title: Ex Vivo Test of New Stroke Treatment Using Magnetic Nanorobots
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, ZHANG Li, Professor, Chinese University of Hong Kong
Other Study IDs: 2020.384
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tissue plasminogen activator (tPA) is the FDA approved thrombolytic drug for patients with acute ischemic stroke. While transcatheter endovascular therapy is widely accepted as an effective method for targeted blood vessels via a catheter to elicit ischemic necrosis.

To improve targeting accuracy administrated tPA and avoiding collateral tissue damage, we developed a magnetic nanorobotic system to active system to active intravenous delivery of tPA for targeted thrombus removal. Here human placenta will be used as an ex vivo model for human cerebral vascular system in our ex vivo thrombolysis study. Our magnetic nanorobotic system encapsulated with tPA overcomes the limitations of passive thrombolytic therapy with tPA alone and will be a promising approach for the treatment of ischemic stroke and other thrombotic diseases

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women at 20-45 years of age of any ethic origin, giving childbirth with natural delivery or caesarean sections after 37-42 weeks of gestation.
* Healthy singleton pregnancy.
* Participant able to give voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

* Abnormal prenatal development (e.g intrauterine growth restriction)
* Early preterm birth < 37 weeks
* Verbal Confirmation of hypercholesterolemia
* Family history of stroke or vascular disease
* Type I or Type II diabetes and gestational diabetes
* Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative.
* Clinically significant abnormal laboratory results at screening.
* Any other active or unstable medical condition.
* History of liver disease.
* History of hypertension (including pre-eclampsia)

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Healthy pregnant women at 20-45 years of age of any ethic origin, giving childbirth with natural delivery or caesarean sections after 37-42 weeks of gestation.
  * Healthy singleton pregnancy.
  * Participant able to give voluntary, written, informed consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Thrombolysis performance | 1 -2 hours
  Size of thrombus by angiography, mm
Time for recanalization | 1 -2 hours
  Time for recanalization of occluded vessels, mins
Damage to vessels | 1 -2 hours
  Histological damage evaluation. The vessels are sectioned and stained with H&E stain

SECONDARY OUTCOMES:
Stability of magnetic nanorobots | 1 - 2 hours
  Controllability of the magnetic nanorobots. The loss in mass of nanorobots after magetic navigation in blood vessels is measured.
Dosage requirement | 1 - 2 hours
  Dosage requirement of nanorobots and thus t-PA, mg
Distribution of administrated nanorobots | 1 - 2 hours
  The distribution of administrated nanorobots. The position of nanorobots is tracked by MRI.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Advanced Nanomaterials & Microrobotics Laboratory, Room 202, William M.W Mong Engineering Building, CUHK and Room 508, Li Ka Shing Medical Sciences Building, Prince of Wales Hospital, Shatin, New Territories
  - Department of Obstetrics and Gynaecology, Prince of Wales Hospital, Shatin, New Territories

IPD SHARING:
Plan to Share IPD: No